CLINICAL TRIAL: NCT04039750
Title: Use of Antibiotic Irrigation to Decrease Wound Infections in Pediatric Perforated Appendicitis
Acronym: PA protocol
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00088360
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Perforated Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Suction; Clindamycin; Gentamicins

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 1 of 2 groups. Group "A" will be Antibiotic Irrigation with suction and Group "B" will be Suction Alone.
Who Masked: Participant
Masking Description: there is no masking after randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic irrigation with suction (Experimental): Group A: You will receive antibiotic irrigation with suction if a PA is found during surgery
  Interventions: Drug: antibiotic rinse with suction
- suction only (Active Comparator): Group B: You will receive suction alone if a PA is found during surgery
  Interventions: Procedure: suction only

INTERVENTIONS:
Drug: antibiotic rinse with suction — antibiotic rinse with suction
  Other Names: Clindamycin, gentamycin
  Arms: Antibiotic irrigation with suction
Procedure: suction only — no irrigation, suction only
  Arms: suction only

SUMMARY:
The proposed study will investigate whether antibiotic irrigation using a gentamicin/clindamycin solution during laparoscopic appendectomy is superior in preventing postoperative wound infections and IAA in perforated appendicitis compared to suction without irrigation. This will be the first prospective study to compare these two options in pediatric PA.

DETAILED DESCRIPTION:
This study is for pediatric patients who are having an appendectomy and have a perforated appendix. The purpose of this study is to see whether antibiotic irrigation using gentamicin, clindamycin and suction during the surgery works better when compared to suction alone when cleaning the stomach cavity.

Arm A patients will have their abdomen irrigated with the antibiotics, gentamycin and clindamycin, and then the wound will be suctioned out. Arm B patients will not have the antibiotic irrigation but will have their wound suctioned.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or younger
2. Scheduled to undergo laparoscopic appendectomy
3. Preoperative or intra-operative diagnosis of perforated appendicitis (PA).
4. Willingness to undergo treatments, provide written informed consent, and participate in follow-up.

Exclusion Criteria:

1. Male or female older than 18 years of age
2. Declined to undergo laparoscopic appendectomy
3. Not willing to provide written informed consent or undergo randomization of treatment
4. Pregnancy

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
wound complications | 30 days
  The overall objective is to change the postoperative wound complications and IAA after laparoscopic appendectomy for perforated appendicitis in pediatric patients. The outcome will be measured by tracking any wound complications that these patients have and comparing the incidence between treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gates, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health - Upstate, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No